CLINICAL TRIAL: NCT04446806
Title: A Prospective Single Center Study of Prevention and Treatment of Differentiation Syndrome in Patients With Acute Promyelocytic Leukemia
Brief Title: Prevention and Treatment of Differentiation Syndrome in Patients With Acute Promyelocytic Leukemia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: APL-01
Record Dates: First submitted 2020-03-29; First posted 2020-06-25 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-03

CONDITIONS: Safety and Efficacy
MeSH Terms: interventions — ruxolitinib

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Ruxolitinib — Ruxolitinib as second treatment in patients with severe DS failed in responding to hormone.Furthermore

SUMMARY:
With the introduction of all-trans-retinoic acid (ATRA) and arsenic,the outcome of patients with acute promyelocytic leukemia (APL)has been improved considerably over the last decades.However，early deaths (EDs), mainly due to APL-specific coagulopathy, differentiation syndrome (DS)emerge as a major threat to APL patients.We observe and evaluate the effectivity of induction therapy in patients with APL. Administrate intravenous dexamethasone to prevent or preemptive treat DS. Assess the efficacy and safety of ruxolitinib as second treatment in patients with severe DS with no respond to dexamethasone.Furthermore，the changes of spectrum of cytokines are monitered to find the relationship between the cytokines and the severity of DS.

DETAILED DESCRIPTION:
Adults ages 18-75 with primary acute promyelocytic leukemia.

Design:

The induction therapy with ATRA 25mg/m2/d and ATO 10mg/kg/d should be started as soon as the diagnosis of APL confirmed.

Intravenous dexamethasone at a dose of 5-20 mg daily must be started if the WBC count greater than 5e+9/L (before or during the treatment with ATRA) as prevention or preemptive therapy of DS.

Idarubicin (4-10 mg/m2 /d*3d) and hydroxyurea（1.0-3.0g/d）can be given as leukocyte lowering therapy which may lessen the risk of DS.

When the progression of clinical symptoms of DS with no response to dexamethasone,ATRA must be stopped and ruxolitinib (5-20mg /d) should be administrated to reduce the production of cytokines.

Participants should stay in the hospital during the treatment for about 4 weeks.

The changes of spectrum of cytokines are monitored to discover the potential relationship between the cytokines and the severity of DS.

Participants will visit every 1 months after CR for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of primary acute promyelocytic leukemia.
* ECOG score≤3.
* Must be able to understand and willing to participate in the study and sign the informed consent.

Exclusion Criteria:

* Refractory/secondary acute promyelocytic leukemia.
* Severe complications such as myocardial infarction, chronic cardiac insufficiency, hepatic failure, renal insufficiency, etc.
* Clinically uncontrolled active infections.
* Malignant tumors with other progresses.
* Ecg: QT interval > 450 ms.
* Allergic to arsenic agent.
* Pregnant or lactating women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
complete remission rate | during the induction treatment
  complete remission rate after treated by the induction regimen with ATRA and Arsenite
incidence and severity of differentiation syndrome | during the induction treatment
  All symptoms and signs associated to DS should be paid closely attention to.

SECONDARY OUTCOMES:
overall survival | from the day of first patient treatment up to 36 months after the last patient's enrollment
  from the date of inclusion to date of death, irrespective of cause

CONTACTS AND LOCATIONS:
Overall Officials: Qian Wu, Study Chair — First Affiliated Hospital, Soochow University Suzhou, Jiangsu, China, 215000
Locations (1):
- First Affiliated Hospital, Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No